CLINICAL TRIAL: NCT04976556
Title: Breast Carcinoma Detection in Ex-vivo Fresh Breast Surgical Specimens Using the Histolog Scanner, Slide-free Confocal Microscopy Scanner
Brief Title: Breast Cancer Detection in Breast Surgical Specimens With the Histolog Scanner, Slide-free Confocal Microscope
Acronym: Hibiscuss
Status: Completed | Type: Observational
Sponsor: SamanTree Medical SA (Industry)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: Hibiscuss
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Confocal Microscopy; Fresh Tissue Imaging; Intraoperative Assessment; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Histolog Scanner — imaging of fresh lumpectomy specimens with the Histolog Scanner, confocal microscopy scanning medical imaging device

SUMMARY:
Study to assess the capability of physicians (breast surgeons and pathologists) to recognize breast cancer in images of fresh lumpectomies generated with the Histolog Scanner, a recent large field-of-view confocal laser scanning medical imaging device.

DETAILED DESCRIPTION:
Breast cancer is the commonest cancer in female worldwide and breast-conserving surgery (BCS) became the most frequently performed surgical treatment for women with early-stage breast cancer. The ability to identify subclinical and deep-seated tumor during BCS is still difficult, and the surgeon must rely on nonspecific visual changes and manual palpation of subtle irregularities to guide cancer excision. Although there is no consensus on negative surgical margins, at least 20 % of patients undergo more than one procedure to achieve acceptable margins as part of breast-conserving strategy. The development of reliable intraoperative assessment tools which can provide a timely indication of whether re-excision in tumor bed after BCS is indicated at the time of primary surgery would be an asset. The Histolog Scanner is a recent confocal microscope designed for fresh tissue ex-vivo medical imaging with high resolution and speed to guide intraoperative assessment and offer support in clinical decision making. Allowing the quickest and most effective intraoperative assessment of breast surgical specimen regardless of center clinical workflow and intraoperative availability of pathologist, is the aim of this international study. The main objective is to demonstrate that both pathologists and surgeons are able to detect breast cancer tissues in Histolog Scanner images of breast surgical specimens.

Fresh Breast surgical specimens with breast cancer (invasive or in-situ) will be imaged with the Histolog Scanner prior Standard-of-Care final assessment in pathology. Content of the images will be reviewed by a board of expert pathologists using the gold standard (H&E-stained images) as reference. Blind assessment of the breast cancer content of these Histolog Scanner images will be realized by breast surgeons and pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient ≥18 years old
* Women with diagnosed, operable invasive or in situ ductal carcinoma, invasive lobular carcinoma who are deemed breast surgery candidates (i.e. lumpectomy or mastectomy).
* Patient able to read, understand and give informed consent

Exclusion Criteria:

* Patient not informed
* Patient previously treated for breast carcinoma
* Patient has undergone presurgical neo-adjuvant treatment
* Patient is pregnant/lactating
* Patient is male
* Participation in any other clinical study that would affect data acquisition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient are selected by breast surgeons during their standard-of-care preoperative consultations
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy, Sensitivity, Specificity, Positive predictive value, Negative predictive value for breast cancer detection | Through study completion, an average of 1 year
  Quantification of the performance achieved by breast surgeons and pathologists for breast cancer detection in Histolog Scanner images

SECONDARY OUTCOMES:
Accuracy for breast cancer diagnosis | Through study completion, an average of 1 year
  Quatification of the performance achieved by pathologists to differentiate breast cancer subtype (IDC, DCIS or ILC) in Histolog scanner images.

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Conversano, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Marie-Christine Mathieu, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Conversano A, Abbaci M, van Diest P, Roulot A, Falco G, Ferchiou M, Coiro S, Richir M, Genolet PM, Clement C, Casiraghi O, Lahkdar AB, Labaied N, Ragazzi M, Mathieu MC. Breast carcinoma detection in ex vivo fresh human breast surgical specimens using a fast slide-free confocal microscopy scanner: HIBISCUSS project. BJS Open. 2023 May 5;7(3):zrad046. doi: 10.1093/bjsopen/zrad046. PMID 37178160